CLINICAL TRIAL: NCT00652444
Title: Effect Of Ezetimibe Coadministration With Simvastatin In A Middle Eastern Population: A Prospective, Multicentre, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Effect Of Ezetimibe Coadministration With Simvastatin In A Middle Eastern Population: A Prospective, Multicentre, Randomized, Double-Blind, Placebo-Controlled Trial (0653-151)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653-151; 2008_004
Record Dates: First submitted 2008-03-31; First posted 2008-04-03 (Estimated); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Coadministration arm: simvastatin 20mg and ezetimibe 10mg
  Interventions: Drug: ezetimibe; Drug: simvastatin
- 2 (Experimental): Monotherapy arm: simvastatin 20mg and ezetimibe placebo
  Interventions: Drug: simvastatin; Drug: Placebo (Unspecified)

INTERVENTIONS:
Drug: ezetimibe — ezetimibe 10mg. Blood samples were collected again at the end of study treatment, week 6.
  Other Names: Zetia®; EZETROL®; MK0653
  Arms: 1
Drug: simvastatin — simvastatin 20mg . Blood samples were collected again at the end of study treatment, week 6.
  Other Names: Zocor®; MK0733
Drug: Placebo (Unspecified) — Matching ezetimibe placebo
  Arms: 2

SUMMARY:
The primary outcome was percentage reduction of LDL-C after 6 weeks of randomization.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known Coronary Artery Disease (CAD) and primary hypercholesterolemia, who are being treated with simvastatin 20mg. Simvastatin consumption meant that subjects must be currently taking simvastatin 20mg daily, and by history have taken at least 80% of daily evening doses for the preceding 6 weeks prior to baseline visit
* Age of at least 18 years and 75 years or less
* Calculated LDL-C concentration of at least 2.6 and 4.1mmol/l or less using the Friedewald equation, and triglyceride of less than 3.99 mmol/l

Exclusion Criteria:

* Congestive heart failure (defined as New York Heart Association class III or IV heart failure)
* Uncontrolled cardiac arrhythmias
* Acute coronary syndrome, coronary bypass surgery or coronary angioplasty within 3 months of study entry
* History of unstable or severe peripheral artery disease within 3 months of study entry
* Uncontrolled hypertension at study entry
* Uncontrolled or newly diagnosed diabetes mellitus (within 3 months of study entry)
* Uncontrolled endocrine or metabolic diseases known to influence serum lipids and lipoproteins; known impairment of renal function
* Active or chronic hepatic and hepatobiliary disease
* Disorders that would limit study evaluation or participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2003-09; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Percentage reduction of LDL-C after 6 weeks of treatment. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Zubaid M, Shakir DK, Bazargani N, Binbrek A, Gopal R, Al-Tamimi O, Bakir S. Effect of ezetimibe coadministration with simvastatin in a Middle Eastern population: a prospective, multicentre, randomized, double-blind, placebo-controlled trial. J Cardiovasc Med (Hagerstown). 2008 Jul;9(7):688-93. doi: 10.2459/JCM.0b013e3282f3a1b1. PMID 18545068